CLINICAL TRIAL: NCT02414542
Title: A Multicentre, Prospective, Observational Clinical Study Evaluating the Outcomes of a Cementless Metaphyseal Short Stem After Hip Arthroplasty
Brief Title: Minima Clinical Study
Status: Completed | Type: Observational
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: H-11
Record Dates: First submitted 2015-03-31; First posted 2015-04-10 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Total Hip Arthroplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MINIMA stem

SUMMARY:
Post-marketing clinical study,international, multi-centre, prospective, observational. The investigation will be carried out in 2 sites in Europe for a maximum total number of 160 patients.The aim of this study is to assess clinical, radiographic and subjective outcomes after hip arthroplasty with a cementless metaphyseal MINIMA short stem, define the survivorship of the implant and identify possible risk factors that may lead to failure.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders
2. Age ≥ 18 years old
3. Life expectancy over 5 years
4. Any race
5. Ambulatory patients
6. Painful primary coxarthrosis
7. Painful secondary coxarthrosis
8. Avascular necrosis
9. Willingness to comply with rehabilitation and study evaluation and ability to return for follow-up visits
10. Signed study-specific Informed Consent Form

Exclusion Criteria:

1. Body mass index over 28 kg/m2 for the modular version
2. Requiring revision of previous standard femoral stem
3. Symptomatic OA of the knees, spine, ankles or contralateral hip, if it can interfere with the evaluation of the target hip according to the Investigator
4. Previous hip replacement (resurfacing or THR) on the contralateral side and whose outcome is achieving an HHS< 60 points
5. Significant proven or suspicious infection of the target hip
6. Any serious infectious disease before the study according to the Investigator
7. Muscular insufficiency that may compromise functional recovery
8. Proven osteopenia and osteoporosis severe enough to compromise the stem support according to the Investigator
9. Known or suspicious hypersensitivity to the metal of the implant
10. Recurrent medical history of immune-mediated reactions or other systemic immune disorders
11. Vascular insufficiency or peripheral neuropathy of lower limbs severe enough to interfere with the study evaluation according to the Investigator
12. Current treatment or treatment for any malignancy within the previous 2 years before the preoperative visit
13. Previous organ transplant
14. Any intercurrent chronic disease or condition that may interfere with the completion of the 60-month follow-up, such as liver disease, severe coronary disease, or other clinically significant condition that the Investigator feels may affect the study evaluation
15. Known co-existent medical condition where death is anticipated within five years due to the pre-existing medical condition
16. Any clinically significant finding that would place the patient at health risk, impact the study, or affect the completion of the study
17. Current alcoholism, and/or any known current addiction to pain medications or drugs
18. Any psychiatric illness that would prevent comprehension of the details and nature of the study
19. Participation in any experimental drug/device study within the 6 months prior to the preoperative visit
20. Unwillingness or inability to comply with rehabilitation and to return for follow-up visits
21. Women of childbearing potential who are pregnant, nursing, or planning to become pregnant, and those who do not agree to remain on an acceptable method of birth control throughout the entire study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected for recruitment into the study from the general diagnosis population of patients requiring a primary hip arthroplasty, due to symptomatic painful degenerative joint diseases (NDJD). Patients requiring a revision of a previous failed stem cannot be enrolled into the clinical evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-09; Primary Completion 2017-12 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score (HHS) | 24 months
UCLA activity score | 24 months
Time up and go test (TUG) | 24 months
Range of motion (ROM) | 24 months

SECONDARY OUTCOMES:
Hip disability and Osteoarthritis Outcome Score (HOOS) | 24 months
Implant stability measured by radiographic evaluations | 24 months
Revision rate | 24 months
Incidence of device-related Adverse Events/Serious Adverse Events | 24 months

OTHER OUTCOMES:
Mid-term clinical outcomes: Harris Hip Score and Hip disability and Osteoarthritis Outcome Score (HOOS) | 60 months
Incidence of device-related Adverse Events and Serious Adverse Events | 60 months
Survival rate (Kaplan Meier) | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Zagra, Principal Investigator — I.R.C.C.S. Galeazzi
Locations (1):
- I.R.C.C.S. Galeazzi, Milan, Italy